CLINICAL TRIAL: NCT02791542
Title: Sorting and Expression Profiling of Airway Cells From Humans (The SEARCH Study)
Acronym: SEARCH
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 16-18550; R01HL138424 (NIH); U19AI077439 (NIH)
Record Dates: First submitted 2016-06-01; First posted 2016-06-06 (Estimated); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bronchial brushes and lavage Sputum, induced Whole blood Urine Serum Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Asthma: Participants with a history of asthma
- Healthy controls: Participants without a history of asthma
- Asthma Bronchoscopy sub-group: Participants with a history of asthma who will undergo the same procedures as other healthy controls with the addition of bronchoscopy
- Healthy Bronchoscopy sub-group: Participants without a history of asthma who will undergo the same procedures as other healthy controls with the addition of bronchoscopy

SUMMARY:
This will be a single site, mechanistic study of asthmatic subjects and healthy, non-asthmatic controls involving a baseline characterization visit and a research bronchoscopy visit. We will identify differences in airway epithelial epigenetic enhancer signatures in asthma, by analyzing freshly isolated airway epithelial cells from healthy controls and from well-characterized subjects with asthma.

DETAILED DESCRIPTION:
The airway epithelium is critical for normal lung function and changes in the epithelium are central to the development of asthma. Precise regulation of gene transcription is essential for airway epithelial cell differentiation and transcription changes lead to many abnormalities seen in asthma. Despite the dominant role of enhancers in regulating transcription, little is known about how these DNA regulatory elements control airway epithelial cell transcription or about how enhancer activity differs in asthma compared to health. Closing this knowledge gap will have a major impact on our understanding of normal epithelial development and asthma. In addition, enhancer-based approaches for reprogramming the airway epithelium promise to be powerful tools for dissecting mechanism that will set the stage for developing a new class of precisely targeted treatments for asthma. Our overall goals are to identify enhancers that are important in regulation of key airway epithelial cell genes, to determine how enhancer activity changes in asthma, and to develop approaches for targeting the activity of these enhancers.

ELIGIBILITY:
Inclusion Criteria (Healthy participants):

1. Male and female subjects between the ages of 18 and 70 years
2. Ability to provide written informed consent and ability to comply with the requirements of the study
3. No hyperreactivity to methacholine (PC20 FEV1 Methacholine >16 mg/mL)
4. No history of allergic rhinitis/seasonal allergies

Inclusion Criteria (Asthmatic participants):

1. Male and female subjects between the ages of 18 and 70 years
2. Ability to provide written informed consent and ability to comply with the requirements of the study
3. History of asthma
4. No use of oral or inhaled corticosteroids for the treatment of asthma during the past 6 weeks
5. Hyperreactivity to methacholine (PC20 FEV1 Methacholine < 8 mg/ml)

Exclusion Criteria:

The same exclusion criteria will apply to both Sub-studies.

1. Current smokers, defined by (a) >5 cigarettes smoked in past 12 months, and (b) ≤ 8 weeks since last time smoking; or former smokers who have a total smoking history ≥10 pack-years
2. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
3. Subjects with a history of lung disease other than asthma
4. Subjects with a history of a medical disease, which in the opinion of the Investigator may put the subject at extra risk from study-related procedures or because the disease may influence the results of the study
5. Prior esophageal hernia surgery.
6. Current participation in an investigational drug trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and asthmatic participants recruited from community advertising
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Measure the genomic location of enhancers in genes previously found to be differentially expressed in asthma vs health using H3K27ac ChIP-seq and ATAC-seq on airway epithelial brushings. | Between 1-12 weeks
  We previously identified changes in epithelial gene expression in individuals with asthma. To identify candidate enhancers that account for these changes, we will use Drop-seq, ChIPseq and ATAC-seq to analyze freshly isolated airway epithelial cells from healthy controls and from well-characterized subjects with asthma.
Assessment of persistence of signatures of airway inflammation | 1-12 weeks and at 10-14 months
  Perform epithelial brush gene expression profiling and sputum induction on longitudinal samples obtained at 12 months after the initial bronchoscopy, to assess stability of type-2 and non-type-2 pathways that are dysregulated in asthma. (Achieved via the PISA sub-study)

SECONDARY OUTCOMES:
Measure gene expression by RNA sequencing in both airway brushes and BAL cells for assessment of non-type-2 pathways differentially expressed in asthma vs health. | Between 1-12 weeks
  Perform bronchoalveolar lavage (BAL) cell flow cytometry and epithelial brush gene expression profiling to look for non-type-2 pathways that are dysregulated in asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Bhakta, MD, PhD, Principal Investigator — University of California, San Francisco; Prescott Woodruff, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No